CLINICAL TRIAL: NCT02987803
Title: Helping Mothers Select Better Childbirth Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Neel Shah, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB16-1371
Record Dates: First submitted 2016-11-17; First posted 2016-12-09 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Cesarean Section
Keywords: Patient Engagement; Public Reporting; Quality Measurement
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants in the control group will receive educational articles about obstetric hospitals. The articles will prompt the participant to look up hospitals in their geographic location. Participants will not know they are participating in a trial.
- Data Group (Experimental): Participants in the intervention group will receive an educational module designed to support them in selecting a delivering hospital, which will include an educational video, articles, and a data tool with cesarean delivery rate data for hospitals in their geographic location.
  Participants will not know they are participating in a trial.
  Interventions: Other: Data

INTERVENTIONS:
Other: Data — The tool displays star ratings of hospitals on how labor-friendly they are. The star ratings (1 through 5) are based on hospital-level cesarean delivery rates. The data comes from The Leapfrog Group and is supplemented by publicly available state data. The data displayed will be customized to the users geographic location.
  Arms: Data Group

SUMMARY:
The investigators aim to conduct a randomized controlled trial of women who are pregnant or considering pregnancy to understand whether women provided with specific data on hospital-level cesarean delivery rates are more likely to select higher quality hospitals, defined as hospitals with cesarean delivery rates below the Federal HealthyPeople 2020 target of 23.9%.

DETAILED DESCRIPTION:
The choice of a childbirth provider is one of the most consequential decisions a pregnant woman makes. The hospital she delivers at is a better predictor of many treatment decisions than her own risks or preferences. For example, choosing the wrong hospital can increase the risk of cesarean delivery up to 10-fold. Cumulatively, avoidable cesarean deliveries are estimated to cause 20,000 major surgical complications, $5 billion in spending, and unmeasured pain each year in the United States.

The proposed project aims to prevent these harms by empowering women to choose hospitals with risk-appropriate cesarean delivery rates. Preliminary research indicates that the majority of women may not understand how hospital-level quality data applies to them personally. In a test sample of 1,000 demographically diverse pregnant mothers, over half do not know if hospital-level cesarean delivery rates are important, and the overwhelming majority do not know if obstetrical infection rates, maternal or neonatal birth trauma rates, or hospital quality metrics are important when selecting their hospital. The investigators will conduct a randomized controlled trial of women using Ovia Health mobile applications to track their fertility or pregnancy to understand whether women provided with location-specific cesarean delivery rate data along with education about the importance of hospital-level cesarean delivery rates are more likely to select higher quality hospitals than women provided with education alone.

The study is labeled double blind, but the investigators recognize uncertainty on this framework. Though subjects will be exposed to different information they do not know they were in a trial. At the point that outcomes are collected, researchers will not know which group the subject was randomized because outcomes are self-reported.

ELIGIBILITY:
Inclusion Criteria:

* Ovia Fertility users that are trying to conceive and are not infertile or Ovia Pregnancy users within the United States in their first trimester who have NOT chosen a delivery hospital or provider.

Exclusion Criteria:

* People who do not use Ovia Health mobile applications, Ovia Pregnancy users beyond the first trimester of their pregnancy, Ovia Fertility users that are not infertile (as defined by women under 35 that have been trying for more than 12 months, and women over 35 that have been trying for over 6 months) and Ovia Pregnancy/Fertility users who have selected their delivering hospital or provider.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120621 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Hospital Selection | Up to 12 months
  Enrollees will be asked to self-report the hospital where they delivered. Hospitals will be categorized into a five-star quality rating scale based on the corresponding quintile of their cesarean section rate at the state level, as reported to the Leapfrog Group and other state data sources. Our primary outcome will be the average star rating of hospitals selected by control and intervention group enrollees. We will also report the proportion of enrollees in each group selecting hospitals of each star rating, as well as selecting hospitals that do not report their cesarean section rate.

SECONDARY OUTCOMES:
Knowledge of Hospital-Level Differences | Up to 12 months
  Participants' response to a survey question about thinking there are differences in cesarean delivery rates between hospitals in their community
Hospital Impact on Cesarean Delivery Risk | Up to 12 months
  Participants' response to a survey question about thinking the hospital they choose will impact their chances of having a cesarean delivery
Use of Rates in Hospital Selection | Up to 12 months
  Participants' response to a survey question about looking at cesarean delivery rates when choosing their childbirth hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ateev Mehrotra, MD, MPH, Principal Investigator — Harvard Medical School (HMS and HSDM); Neel Shah, MD, MPP, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehrotra A, Wolfberg A, Shah NT, Plough A, Weiseth A, Blaine AI, Noddin K, Nakamoto CH, Richard JV, Bradley D. Impact of an educational program and decision tool on choice of maternity hospital: the delivery decisions randomized clinical trial. BMC Pregnancy Childbirth. 2022 Oct 10;22(1):759. doi: 10.1186/s12884-022-05087-y. PMID 36217115
- See also: Ariadne Labs — https://www.ariadnelabs.org/
- See also: Ovia Health — https://www.oviahealth.com